CLINICAL TRIAL: NCT03230344
Title: Surgical Periodontal Intervention With Simultaneous Versus Delayed Endodontic Treatment in Concurrent Endodontic-Periodontal Lesion Without Communication - An Interventional Study
Brief Title: Periodontal Surgery With Early vs Delayed Endodontic Treatment in Endo-Perio Lesions Without Communication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ruchika perio
Record Dates: First submitted 2017-07-13; First posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Periodontal and Endodontic Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Periodontal treatment initiated with scaling and root planing along with root canal treatment and followed by open flap debridement after 6 weeks.(Open flap debridement simultaneously with root canal treatment )
  Interventions: Procedure: open flap debridement
- Group 2 (Experimental): Periodontal treatment initiated with scaling and root planing followed by open flap debridement after 6 weeks. Endodontic treatment will be initiated after 3 months of periodontal surgery.(open flap debridement and delayed root canal treatment )
  Interventions: Procedure: open flap debridement

INTERVENTIONS:
Procedure: open flap debridement — open flap debridement simultaneously with root canal treatment
  Other Names: root canal treatment
  Arms: Group 1
Procedure: open flap debridement — open flap debridement and delayed root canal treatment
  Other Names: root canal treatment
  Arms: Group 2

SUMMARY:
The aim of this study is to evaluate the periodontal parameters in terms of periodontal healing by periodontal surgical therapy with simultaneous or delayed endodontic therapy in management of concurrent endodontic -periodontal lesion without communication

DETAILED DESCRIPTION:
INTRODUCTION

The term " Endodontic-Periodontal " lesion has been proposed to describe the destructive lesions resulting from inflammatory products found in varying degrees in both the periodontium and the pulpal tissues. The term concurrent endodontic periodontal lesion without communication applies to a tooth that has an infected root canal system with some form of apical periodontitis plus marginal periodontal disease with pocketing but the periapical and periodontal disease do not communicate with each other.

Although there are many factors, the primary cause of both diseases is the presence of bacterial infection with complex microbial flora. Based on microbiological studies many authors have reported the similarity between bacterial flora associated with endodontic and periodontal infections. Therefore periodontal pocket may be a source of bacteria for root canal system or vice versa and cross seeding of bacteria can occur in either direction through communication pathways. An untreated infection of one of these tissues can lead to signs or symptoms of disease within the other tissue.

Observations based upon review articles and case reports has suggested, if the root canal system is infected, endodontic treatment should be commenced prior to any periodontal therapy in order to remove the intra-canal infection before any cementum is removed in case of concurrent endodontic - periodontal lesions without communication. Treatment results of endodontic therapy should be evaluated in 2-3 months and only then periodontal treatment should be considered.

Concerns about the possibility that endodontically treated teeth might not respond to periodontal therapy are certainly not new. Histological examination of human teeth concluded that endodontic therapy had adversely affected periodontal healing. Teeth that had undergone endodontic therapy did not respond well to regenerative procedures as teeth that had not undergone such treatment. It has been advocated to perform periodontal therapy before endodontic obturation because of the concern that the leakage of endodontic sealer would hinder repair, regeneration or both. There is a negative impact of certain root canal filling materials on fibroblast attachment to the dentin surface of extracted third molars. Also endodontic therapy performed simultaneously with or soon after periodontal surgery adversely affected the formation of new bone, new cementum and new attachment. It was also found in a study that periapical pathology was not significantly correlated to mean pocket depth reduction after non surgical and surgical treatment of horizontal and vertical defects .

The microflora in infected root canals of teeth that have concurrent endodontic and periodontal diseases is more complex than in teeth with infection confined to the periapical region.

All the above findings are based on microbiological, histological, case-reports, retrospective and in vitro studies, management of concurrent endodontic periodontal lesions need more evidence based investigations. So far no clinical study has compared periodontal healing along with or without endodontic therapy. It is hypothesized that endodontic treatment did not influence the periodontal outcomes after periodontal surgery in endodontic-periodontal lesion without communication.

Thus the aim of our study is to evaluate the periodontal parameters in terms of periodontal healing by periodontal surgical therapy with simultaneous or delayed endodontic therapy in management of concurrent endodontic -periodontal lesion without communication.

MATERIAL AND METHOD

This study will be conducted in Department of Periodontics and Oral Implantology in collaboration with Department of Conservative Dentistry and Endodontics, Post Graduate Institute of Dental Sciences , Rohtak.

STUDY POPULATION Patients will be recruited from regular out patient department of the Department of Periodontics and Oral Implantology, Department of Conservative Dentistry & Endodontics and Department of Oral medicine, Diagnosis and Radiology.The study will be conducted as follows:- This Interventional study will include systemically healthy minimum 36 patients with chronic periodontitis having at least one tooth involving endodontic periodontal lesion which will be further divided into two groups (minimum 18 each) based on patient's consent for treatment.

1. Simultaneous endodontic periodontal therapy group (Group 1) Scaling and root planning will be performed simultaneously with non surgical endodontic treatment (in the form of root canal treatment). After 6 weeks of scaling and root planning , periodontal surgery will be performed in the form of open flap debridement.
2. Delayed endodontic therapy group (Group 2) Periodontal treatment initiated with scaling and root planning followed by periodontal surgery in the form of open flap debridement after 6 weeks. Endodontic treatment will be initiated after 3 months of periodontal surgery.

Prior informed consent will be taken from each patient after explaining the procedure in patient's language along with risk and benefits involved.

METHODOLOGY Patients will be allocated to group1 and group 2. The study will be conducted as follows:- Presurgical therapy:- which will be including

i. Oral hygiene instructions ii. Full mouth supragingival and subgingival scaling and root planning with ultrasonic scaler, hand scaler and curettes.

iii. In group 1 conventional root canal therapy will be performed simultaneously to presurgical therapy.

Surgical therapy:- In both groups periodontal surgical procedure in the form of open flap debridement will be performed after 6 weeks of SRP.

A probing stent will be fabricated for every patient,relative to which attachment loss will be measured.

In group 2 conventional root canal therapy will be performed 3 months after periodontal surgical procedure.

CLINICAL PARAMETERS

1. Full mouth indices to be recorded at baseline

   * Bleeding on probing
   * Probing Pocket depth
   * Attachment loss
2. Site specific indices

   * Plaque index
   * Gingival index
   * Probing Pocket depth
   * Relative attachment loss
   * Bleeding on probing
   * Tooth mobility
   * Relative gingival marginal level Using UNC 15 periodontal probe at 6 sites (mesial, distal, median points at buccal and lingual aspects) per tooth.

Customized bite blocks and parallel angle technique will be used to obtain radiographs.

Clinical parameters will be recorded at baseline, at 6 weeks of nonsurgical phase, at 3 months and after 6 months post surgery for Group 1(6 months of periodontal surgery and endodontic treatment) and group 2 (6 months of periodontal surgery and 3 months of root canal treatment).

PERIODONTAL NON SURGICAL PROCEDURE This involves supragingival and subgingival scaling and root planning to be performed with ultrasonic scaler, hand scaler and curette and will be completed in minimum two sessions.

PERIODONTAL SURGICAL PROCEDURE After administration of local anaesthesia, buccal and lingual/palatal intracrevicular incision will be made and mucoperiosteal flaps will be reflected including atleast one tooth ahead and another behind the tooth. Meticulous defect debridement and root planning will be carried out using area specific curettes and scalers with special effort to remove all the granulation tissue. After instrumentation, the root surfaces will be washed with saline solution in attempt to remove any remaining detached fragments from the defect and surgical field. After debridement mucoperiosteal flaps will be repositioned and secured by using 3-0 non absorbable black silk surgical suture. The surgical area will be protected and covered with periodontal dressing and post operative instructions will be given.

-Instructions will be given for gentle brushing with soft brush and reinstructed for proper oral hygiene postoperatively and will be examined weekly for up to 1 month after surgery and again at 3 month.

CONVENTIONAL ENDODONTIC PROCEDURE After achieving local anaesthesia, access opening will be made with the help of round bur. Then the root canal will be thoroughly debrided followed by copious irrigation and subsequently prepared with the help of endo files. After preparation of the canal, calcium hydroxide intracanal medicament will be placed with the help of 27 gauge endodontic syringe for 10 days and access cavity will be sealed with suitable sealer. Obturation will be performed with gutta percha and zinc oxide eugenol based sealer.

-All parameters will be re-evaluated at recall period of 6 weeks, 3 months and 6 months for Group 1 (conventional endodontic periodontal therapy group) and group 2 (delayed endodontic therapy group).

STATISTICAL ANALYSIS

Data recorded will be processed by standard statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

Patients of age 18 years and above, systematically healthy with chronic periodontitis having at least one tooth involving endodontic periodontal lesion without apical communication with following radiographic and clinical features:

* Wide base pocket, deep pocket depth
* Non vital tooth (confirmed by heat test, cold test and electronic pulp test)
* Radiographic periapical alveolar bone destruction and marginal bone loss without apical communication .

Exclusion Criteria

:• Systemic illness known to affect the periodontium or outcome of periodontal therapy.

* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy.
* Patients allergic to medication (local anaesthetic, antibiotics, NSAID).
* Pregnant or lactating mothers.
* Smokers and tobacco chewers.
* Grade 3 mobile teeth.
* Unrestorable tooth.
* Fractured/perforated roots.
* Developing permanent tooth.
* Previously root canal filled.
* History of recent periodontal treatment within 6 months prior to study.
* Teeth with established endodontic periodontal lesions exhibiting <2mm radioopaque bone between the root apex and the periodontal breakdown and with apical communication found during surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
periodontal parameter: CAL | 7.5 months
  Clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: RUCHIKA LATHER, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Publication
Supporting Information: Study Protocol
Time Frame: 1yr 6months
Access Criteria: PGIDS, Rohtak Haryana